CLINICAL TRIAL: NCT06538090
Title: The Early Movers Pilot Intervention: Encouraging Healthy Movement Behaviours in Infants
Brief Title: Early Movers Pilot Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Alberta Health services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Early Movers
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Child Development; Activity, Motor
Keywords: Questionnaires; Semi-structured Interviews
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: All participants will be randomly assigned to group 1 (intervention) or group 2 (control), in a computer generated 1:1 sequence.
Who Masked: Participant
Masking Description: Participants: While the families will not be told explicitly if they have been assigned to the intervention or control group, they may be able to determine their group based on the information regarding movement behaviours they receive/do not receive during their 2 month immunization appointment.
  Research Coordinator: The research coordinator will be aware of the group allocations as they will be in charge of coordinating random assignment and have to schedule other measures based on their specific allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Movers Intervention (Experimental): Participants will receive an educational resource (i.e., hard copy hand-out), access to a digital app with an online toolkit and weekly text messages that includes tips and supportive messaging.
  Interventions: Behavioral: Early Movers
- Control (No Intervention): Participant will receive standard care.

INTERVENTIONS:
Behavioral: Early Movers — The intervention includes: 1) an educational resource (i.e., hard-copy handout) developed for this study on the 24-Hour Movement Guidelines provided to parents at 2-month immunization appointments by public health nurses, who will answer any questions, followed by a discussion with research staff. 2) Follow-up support via access to a digital app with evidence-based information and support through an online toolkit, an anonymous forum, as well as weekly text messages that include tips and supportive messaging related to the guidelines.
  Arms: Early Movers Intervention

SUMMARY:
Our Early Movers longitudinal study found that adherence to the Canadian 24-Hour Movement Guidelines in infancy is low across demographic groups, impacting overall development. Early Movers is a parent-focused intervention designed to increase dissemination and activation of the 24-Hour Movement Behaviour Guidelines for the Early Years. It adapts an established Australian intervention called INFANT. An important first step is conducting a pilot study.

DETAILED DESCRIPTION:
Our goal is to examine the feasibility and acceptability of the Early Movers intervention, a scalable, theory-based, parent-focused intervention designed to increase dissemination and activation of the 24-Hour Movement Behaviour Guidelines for the Early Years.

Primary Objectives:

1. Explore the feasibility of the Early Movers intervention protocol, including recruitment, retention, data collection, and procedures. Specifically, we will examine:

   1. the willingness of first-time parents to enroll and remain in the study,
   2. data collection completion rates, and
   3. the integrity of the protocol components to all work together and run smoothly.
2. Explore the acceptability of the intervention by parents and public health staff.

ELIGIBILITY:
Inclusion Criteria:

-First time parents of infants who are aged 2 months 0 days through 2 months 30 days at baseline.

Exclusion Criteria:

* Parents who do not confidently speak or read English
* Infants who are regularly cared for by an adult other then their parent/guardian for a number of hours per week (e.g. full time child care)
* Infants born preterm (gestational age <37 weeks)
* Infants born underweight (<2500 g)
* Infants with a medical condition or health complication since birth that could impact their movement behaviours and/or development

Ages: 2 Months to 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2024-10-28 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Feasibility (recruitment) | At recruitment completion, approximately 6 months from the start of recruitment
  How many appointments the research coordinator attends, how many families the research coordinator speaks to, how many families are eligible, and how many families enroll in the trial.
Feasibility (retention) | At data collection completion, approximately 10 months from the start of recruitment
  How many participants drop out
Feasibility (procedures; field observations) | Throughout the 6 months of recruitment
  Field observations recorded by the research coordinator while at public health centres
Feasibility (procedures, interviews) | At recruitment completion, approximately 6 months from the start of recruitment
  Brief semi-structured interviews with public health staff
Feasibility (procedures, interviews) | 4-month follow-up (Infant age: 6 months)
  Brief semi-structured interviews with parents from the intervention group only
Feasibility (data collection) | Baseline (Infant age: 2 months), 2-month follow-up (Infant age: 4 months), 4-month follow (Infant age: 6 months)
  Completion rates of movement behaviour and development measures assessed in the questionnaire
Parent acceptability (interviews) | 4-month follow-up (Infant age: 6 months)
  Brief semi-structured interviews with parents from the intervention group only
Parent acceptability (questionnaire) | 4-month follow-up (Infant age: 6 months)
  Intervention usefulness, satisfaction (content and delivery), and novelty assessed via a parental questionnaire in the intervention group only. This scale includes 4 items with values of 1-5; higher values mean more acceptability
Parent acceptability (app usage) | Between baseline (Infant age: 2 months) and 4-month follow-up (Infant age: 6 months)
  App usage will be tracked in the intervention group only
Public health staff acceptability (interviews) | At recruitment completion, approximately 6 months from the start of recruitment
  Brief semi-structured interviews with public health staff

SECONDARY OUTCOMES:
Physical activity | Baseline (Infant age: 2 months), 2-month follow-up (Infant age: 4 months), 4-month follow (Infant age: 6 months)
  Tummy time measured in a parental questionnaire
Sedentary behaviour | Baseline (Infant age: 2 months), 2-month follow-up (Infant age: 4 months), 4-month follow (Infant age: 6 months)
  Screen time, back time, reading time, restrained time in a stroller, car seat, etc. measured in a parental questionnaire
Sleep | Baseline (Infant age: 2 months), 2-month follow-up (Infant age: 4 months), 4-month follow (Infant age: 6 months)
  Sleep measured in a parental questionnaire
Development | Baseline (Infant age: 2 months), 2-month follow-up (Infant age: 4 months), 4-month follow (Infant age: 6 months)
  Development will be measured with the Ages and Stages Questionnaire (ASQ-3)

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Carson, PhD, Principal Investigator — University of Alberta; Sam Liu, PhD, Principal Investigator — University of Victoria; Kylie Hesketh, PhD, Principal Investigator — Deakin University; Guy Faulkner, PhD, Principal Investigator — University of British Columbia; Lesley Pritchard, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
Due to ethical reasons, individual participant data (IPD) will not be publicly available. De-identified data may be available to other researchers upon reasonable request.